CLINICAL TRIAL: NCT01475422
Title: Effectiveness of the Self Monitoring of Capillary Blood Glucose at Home in Metabolic Control of People With Diabetes Mellitus
Brief Title: Effectiveness of the Self Monitoring of Capillary Blood Glucose at Home
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Vívian Saraiva Veras, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6266936
Record Dates: First submitted 2011-11-10; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conversation Maps Diabetes Education (Experimental)
  Interventions: Behavioral: Conversation Maps Diabetes Education
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Conversation Maps Diabetes Education — The Conversation Maps program is a set of innovative, interactive diabetes education tools developed by the Healthy Interactions, and endorsed by the American Diabetes Association. It consists of four conversation maps covering: 1) how the body and diabetes works, 2) healthy eating and physical activity, 3) treatment with medication and monitoring blood glucose, and 4) reaching the targets with insulin (a fifth map covering gestational diabetes will not be used in this study), and a program manual to help educators successfully implement the program. Participants will be followed for an expected average of 12 weeks.
  Arms: Conversation Maps Diabetes Education
Behavioral: Usual Care — Patients are followed in the medical appointments for evaluation and treatment of diabetes mellitus, according to service routine. Participants will be followed for an expected average of 12 weeks.
  Arms: Usual Care

SUMMARY:
The self-monitoring of capillary blood glucose is part of the package of interventions in diabetes mellitus and an effective therapeutic strategy for the adequate control of the disease; and the continuing education of people with DM is recognized as one of the goals to delay the complications arising from chronic disease and alleviate the symptoms of hypoglycemia and hyperglycemia.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of educational intervention on self-monitoring of capillary blood glucose in metabolic control, knowledge and attitude in two groups of patients with diabetes mellitus: a group of diabetic patients who participate in the Self-Monitoring of Capillary Blood Glucose at Home Program and receive educational interventions (Intervention Group - G1) and a group of diabetic patients who participle in the Self-Monitoring of Capillary Blood Glucose at Home Program and receive conventional treatment (Control Group - G2). As an educational tool in diabetes will be used Conversation Maps which is considered an interactive program of diabetes education.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 Years and older;
* Diagnosis of type 1 and 2 diabetes mellitus;
* In follow-up in the Self-Monitoring of Capillary Blood Glucose at Home Program;
* Have cognitive conditions that enable participation (minimum ability of users to understand issues of data collection instruments, observation of the researcher and/or of the caregivers).

Exclusion Criteria:

* Patients with gestational DM;
* Patients with DM who are not located;
* Those who die in the proposed period for the research;
* Those who dropout the Self-Monitoring of Capillary Blood Glucose at Home Program;
* Those who report difficulties to participate of the study due to work and those with amaurosis;
* Used Conversation Maps as an educational tool.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | baseline, 3 and 6 months post intervention
  Change from baseline in HbA1c at 6 months to less than 7%

SECONDARY OUTCOMES:
Diabetes Knowledge Questionnaire - DKN-A | baseline, 3 and 6 months post intervention
  Change from baseline in DKN-A at six months
Diabetes Attitude Questionnaire - ATT-19 | baseline, 3 and 6 months post intervention
  Change from baseline in ATT-19 at six months

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil